CLINICAL TRIAL: NCT00691587
Title: A Randomized, Double-Blind, Placebo-Controlled Pilot Trial of KB001 in Mechanically-Ventilated Patients Colonized With Pseudomonas Aeruginosa
Brief Title: Pilot Trial of KB001 in Mechanically-Ventilated Patients Colonized With Pseudomonas Aeruginosa
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Humanigen, Inc. (Industry)
Responsible Party: Tillman Pearce, MD, Chief Medical Officer, KaloBios Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KB001-04
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2009-07-31 (Estimated); Status verified 2009-07

CONDITIONS: Pseudomonas Aeruginosa; Ventilator Associated Pneumonia
Keywords: mechanical ventilation; mechanically ventilated; Pseudomonas aeruginosa; ventilator associated pneumonia
MeSH Terms: conditions — Pseudomonas Infections; Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Low-dose KB001, a monoclonal antibody
  Interventions: Biological: KB001
- 2 (Experimental): High-dose KB001, a monoclonal antibody
  Interventions: Biological: KB001
- 3 (Placebo Comparator): Placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: KB001 — Single low-dose, administered intravenously
  Arms: 1
Biological: KB001 — Single high-dose, administered intravenously
  Arms: 2
Biological: Placebo — Placebo single-dose, administered intravenously
  Arms: 3

SUMMARY:
Pseudomonas aeruginosa is an opportunistic pathogen that rarely causes disease in healthy people, but is a significant problem for critically ill or immunocompromised individuals. Experts estimate that there are greater than 100,000 patients in the United States, Europe and Japan where Pseudomonas pneumonia occurs. Patients with Pseudomonas pneumonia currently represent only about 20% of the patients in the hospital who get Pseudomonas infections.

DETAILED DESCRIPTION:
This trial will evaluate KB001 in patients in the intensive care setting who are receiving ventilator therapy and who have Pseudomonas infections. They will receive either placebo, or one of two dose levels of KB001, a Humaneered™, high-affinity antibody fragment that KaloBios is developing for the treatment of Pseudomonas aeruginosa (Pa) infections. This trial will evaluate the ability of KB001 to protect host epithelium and immune cells, and evaluate reduction of pulmonary Pa burden.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent obtained from patient or patient's surrogate if unconscious or altered sensorium
* Age >18 years
* On mechanical ventilation and expected to remain mechanically ventilated for at least 3 days
* Documented pulmonary Pa colonization

Exclusion Criteria:

* Patients with known chronic pulmonary infection with Pa (i.e., patients with cystic fibrosis)
* Patient currently diagnosed with Pa VAP
* Change in systemic antibiotic therapy active against Gram negative bacteria within 72 hours
* Use of an investigational medication within 4 weeks prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
The safety and tolerability of a single dose of KB001. | Day 28

SECONDARY OUTCOMES:
To measure the pharmacodynamic effects of a single-dose of KB001. | Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Jean Chastre, Principal Investigator — Hopital La Pitie Salpetriere
Locations (1):
- Multiple Cities, France